CLINICAL TRIAL: NCT04396743
Title: Comparative Evaluation of Two PRF Formulations on Quality of Life and 2D and 3D Assessment of Healing Outcome of Apicomarginal Defects.
Brief Title: Comparative Evaluation of Two PRF Formulations on Quality of Life and Healing of Apicomarginal Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: vidhiendo
Record Dates: First submitted 2020-04-21; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2019-12

CONDITIONS: Apico Marginal Defects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periapical surgery with placement of prf high clots (Active Comparator): Patients will undergo periapical surgery and PRF-high clot and membrane will be placed inside the bonycrypt and over the denuded root surface respectively before closure of the flap.
  Interventions: Procedure: Periapical surgery with use of prf-high clot and membrane
- Periapical surgery with placement of prf medium clots (Active Comparator): Patients will undergo periapical surgery and PRF-medium clot and membrane will be placed inside the bonycrypt and over the denuded root surface respectively before closure of the flap.
  Interventions: Procedure: Periapical surgery with use of prf-medium clot and membrane

INTERVENTIONS:
Procedure: Periapical surgery with use of prf-high clot and membrane — Periapical surgery will be done followed by placement of prf-high clot into the defect and membrane over the defect before closure of the flap.
  Arms: Periapical surgery with placement of prf high clots
Procedure: Periapical surgery with use of prf-medium clot and membrane — Periapical surgery will be done followed by placement of prf-medium clot in the defect and membrane over the defect before closure of the flap.
  Arms: Periapical surgery with placement of prf medium clots

SUMMARY:
Healing of apicomarginal defects using 2 different formulations of PRF i.e PRF -high and PRF-medium will be assessed and compared using 2D and 3D criteria. Also, in vitro evaluation of the PRF formulations and quality of life will be compared between the two groups.

DETAILED DESCRIPTION:
Periapical surgery is a viable treatment option in teeth with persistent apical periodontitis, especially in cases which fail to heal by non surgical treatment. Kim and Kratchman classified periradicular lesions into categories A-F. Lesions A-C are of endodontic origin without any periodontal pockets and vary with respect to the size of periapical radiolucency while D-F are combined endodontic - periodontal origin and are ranked accoding to the magnitude of periodontal breakdown. Type F defects are commonly referred to as apicomarginal defects and have worst prognosis among all. The lower success rate is attributed to the apical migration of junctional epithelium and intrusion of non osteogenic connective tissue into the periapical region.

Recently, autologous platelet concentrates have been used instead of the conventional practice of using GTR barrier membranes for treating apicomarginal defects. Till date no human study has compared platelet formulations; PRF-high ( 2700 rpm for 12minutes) and PRF-medium (1500 rpm for 14minutes) to see any difference in the bony healing and the quality of life between the two groups and no study have assessed bony healing of the periapical defect with periodontal communication with the use of CBCT.

Thus, the aim of the present study is to investigate the effect of 2 different formulations of PRF on quality of life and healing outcome of periapical defects with periodontal communications . Also, in vitro histological and immunohistochemical evaluation and comparison of the clots prepared from different centrifugation protocols will be done .

ELIGIBILITY:
Inclusion Criteria:

1. Patients of age 16 years and above.
2. Patients with no general medical contraindications for oral surgical procedures (ASA-I and ASA-II according to the classification of the American Society of Anesthesiologist's.
3. periapical defect with periodontal communication.
4. Periodontal pocket >6mm with apicomarginal communication confined to buccal aspect of interproximal space or mid buccal aspect of the root.
5. Negative response to vitality test.
6. failed previous root canal treatment with purulent discharge or failed previous surgery or recurrent episode of purulent discharge.

Exclusion Criteria:

1. Presence of buccal bone on flap elevation.
2. Unrestorable tooth.
3. fractured /perforated roots.
4. smokers.
5. pregnant females and lactating mothers

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2021-04-11 (Estimated); Study Completion 2021-04-11 (Estimated)

PRIMARY OUTCOMES:
Healing of apicomarginal defects. | Baseline to 12 months
  Patients will be checked clinically for absence of signs and symptoms. Radiographic 2D assessment will be done by Rud and Molven criteria as follows:-
  1. Complete healing- defined by re-establishment of the lamina dura
  2. Incomplete healing (scar tissue)
  3. Uncertain healing
  4. Unsatisfactory healing (failure).
  3D healing will be assessed by modified PENN 3D criteria(Schloss et al) as-
  1. Complete healing
  2. Limited healing
  3. Uncertain healing
  4. Unsatisfactory healing.

SECONDARY OUTCOMES:
Assessment of quality of life. | Baseline to day 7 postoperatively
  All patients will be given a questionnaire (Igor Tsesis et al) with 15 questions to evaluate their quality of life for 7 days postsurgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanjay Tewari, Rohtak, Haryana, India